CLINICAL TRIAL: NCT04617990
Title: Knowledge, Attitude and Practice of Physicians Toward The Prescription of Proton Pump Inhibitors in Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ahmad Nassar Ibrahim (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Ahmad Nassar Ibrahim, Ahmed Nassar Ibrahim, Assiut University
Organization: Assiut University (Other)
Other Study IDs: KAP towards PPIs
Record Dates: First submitted 2020-10-31; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to identify the knowledge , attitude and practice toward PPI use among doctors in Egypt

DETAILED DESCRIPTION:
Proton pump inhibitors (PPIs) were developed in the '80s and their use has continuously grown. They represent the first choice in the treatment of acid-related diseases and are currently themost prescribed drugs in the world [1].

In addition, PPIs have become the 8th therapeutic class on the prescription list in 2013. This impacted on health care costs especially in the last decade: in 2010, USA paid $13.9 billion for PPIs [3].

Several studies described a range of adverse events related to longterm PPI use [5,6], some of them are related to increased gastric pH which could alter intestinal bacterial flora and drugs or electrolyteabsorption. Another issue is represented by potential pharmacological interactions between PPIs and other drugs, due to interference with liver metabolic systems, and competition for renal excretion [7-16].

The huge increase in PPI use cannot be justified only by increased prevalence of acid-related diseases or extension of therapeutic indications. Some studies have shown that PPIs are often over-administered in hospital setting, inappropriately prescribed at discharge and maintained by general practitioners (GPs) [1,17,18] A recent research showed that 86% of patients who were prescribed PPIs did not have appropriate indications in the general medical ward of a tertiary Jordanian hospital [2]. Another study showed that PPI were taken by 25.4% of the patients hospitalized in an internal medicine department of a tertiary Greek hospital, but as many as 81.2% of them had no indications [11].

However, the knowledge and practice of physicians in Egypt toward the use of PPI is not well studied.

ELIGIBILITY:
Inclusion Criteria:

1. Physicians dealing with PPI therapy in their specialty including general practitioners, gastroenterologists and non gastroenterologist (hepatologists, otolaryngolists, surgeons, anesthesiologists, pediatriticians and internal medicine physicians.)
2. Who gave consent to participate at the beginning of the questionnaire.

Exclusion Criteria:

* who refuse to gave consent to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Doctors who have completed graduation-MBBCH and have undergone one year internship training but have not yet obtained postgraduate degree.
  2. PhD , M.D. or M.S. or those who have obtained a specialist postgraduate degree.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
five points likert-scale score being | one year
  5 for 'completely agree', 4 for 'almost agree', 3 for 'indifferent', 2 for 'almost disagree', and 1 for 'completely disagree'.